CLINICAL TRIAL: NCT00529646
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Study to Assess the Tolerability, Pharmacokinetics, and Pharmacodynamics of APD791 Administered to Healthy Adult Subjects
Brief Title: Single-Dose Safety Study of APD791 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Christen Anderson, MD, PhD, Arena Pharmaceuticals, Inc.
Allocation: Randomized | Masking: Quadruple
Other Study IDs: APD791-001
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Healthy
Keywords: Healthy adult volunteers
MeSH Terms: interventions — APD791

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: APD791

SUMMARY:
The APD791-001 study is designed primarily to evaluate the safety and tolerability of APD791 when administered as a single oral dose to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, ages 19-45
* Non smokers

Exclusion Criteria:

* History of a bleeding disorder
* Recently donated blood or had significant blood loss
* Current use of a prescription medication
* Pregnant females

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Safety measures to include adverse events, vital signs, 12-lead ECGs, physical examinations, and clinical lab parameters

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic assessments

CONTACTS AND LOCATIONS:
Overall Officials: Christen Anderson, MD, PhD, Principal Investigator — Arena Pharmaceuticals
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- See also: Arena Home Page — http://www.arenapharm.com